CLINICAL TRIAL: NCT06488508
Title: Move-play-explore in Early Childhood Education
Acronym: MoveEarly
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Eivind Aadland, Professor, PhD, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MoveEarly
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Kindergarten Children's Health, Development, Well-being

STUDY DESIGN:
Intervention Model Description: Cluster randomization of 25 kindergartens to the intervention group (professional development) and 25 kindergartens to the control group (standard of care)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Kindergarten staff will participate in 60 hours of professional development over 18 months focused on promotion of movement, play and exploration in the kindergarten setting.
  Interventions: Behavioral: MoveEarly
- Control (No Intervention): Staff receive no professional development and children will receive standard care.

INTERVENTIONS:
Behavioral: MoveEarly — The intervention has two levels: the kindergarten level and the child level.
  1. Staff will receive approximately 60 hours of professional development, including 6 full-day physical seminars, 2 full-day kindergarten visits, 6 written tasks with follow-up webinars and an online resource. The focus will be how to promote movement, play and exploration among children aged 1-6 years.
  2. Staff is supposed to promote children's movement, play and exploration through 7 pedagogical principles: 1. Value, understand and promote movement, 2. Value, understand and promote play, 3. Value, understand and promote exploration, 4. Create rich physical environments, 5. Create opportunities for meaningful participation, 6. Create good balance between challenge and support, and 7. Create good dialogue through action and words.
  Arms: Intervention

SUMMARY:
Evidence is lacking about scalable, effective and sustainable interventions to increase whole-child development in young children. Targeting worrisome trends in physical inactivity and schoolification negatively affecting young children, we will conduct a large cluster randomized controlled trial investigating the effects of professional development of kindergarten staff on kindergarten pedagogical practices regarding movement, play and exploration and child health and development over 18 months. The aim is to recruit 50 kindergartens and 500 children aged 4 years in one county in the western part of Norway to allow for detecting small to moderate effect sizes and ensuring a heterogeneous sample of kindergartens for the study of implementation. Children's physical, mental and socio-emotional development, as well as intervention implementation, will be investigated. The intervention will be developed with strong user involvement from kindergartens and relevant stakeholders to facilitate the development of sustainable solutions.

DETAILED DESCRIPTION:
There are growing concerns about low physical activity levels among young children and schoolification of the kindergartens sector. As 97% of 3-5-year-olds in Norway attend kindergarten, the kindergarten is a unique arena for intervention, laying the foundation for equitable development of health, learning and life opportunities. Yet, evidence of scalable, effective and sustainable interventions to increase physical activity and whole-child development among young children is lacking.

In MoveEarly, we will develop and test a pedagogical intervention focusing movement, play and exploration to counteract trends of increased physical inactivity and instructional teaching practices. For such an intervention to be sustainable, kindergarten staff must lead the implementation of the pedagogical innovation. Thus, we will develop theory on move-play-explore as core elements of a child-responsive pedagogy, investigate how this pedagogy affect child developmental outcomes, develop knowledge on how professional development/continuing education can be co-created among researchers and kindergartens staff, and how such an intervention can be effectively implemented in the kindergarten sector.

Two main research questions will be tested using both quantitative and qualitative methods, applied to both the child and organizational levels:

1. How does the MoveEarly intervention impact children's movement competence, creativity, physical activity, physical fitness, playfulness, explorative behaviour, socio-emotional health, well-being, self-regulation, and early academic learning?
2. How does the MoveEarly intervention interact with different kindergarten contexts to produce various individual and organizational outcomes?

These research questions will be investigated using a cluster RCT with randomization at the kindergarten level, including short- (7-month) and long-term (18-month) follow-ups. The intervention development will include strong involvement from kindergarten owners and staff to provide broad support, buy-in and ownership from kindergarten staff and owners. Thus, we aim to combine a large-scale experimental study with tailored, continuous improvement effort in this sector by taking each kindergarten's contextual factors into account. In this model, to make adaptations within each kindergarten is not considered a lack of fidelity; rather it is a desired process of institutionalization overcoming a common criticism of clinical trials as it increases the value for later scaling and dissemination to the real-world setting. In this way, the aim is to create sustainable solutions for improved child development that can be disseminated in the long-term. Thus, the intervention's development, implementation, and evaluation are framed within a "realist RCT" approach. The intervention model is further framed within a socioecological model, placing the kindergarten as an influential factor for children's health and development.

The intervention has two levels; the kindergarten level and the child level. In response to the challenge of low staff qualifications in general and to implement physical activity specifically, the main component will be an 18-month professional development offered to kindergarten staff. The intervention is structured as a 15-credit continuing education module that provide staff the opportunity to achieve credits for their efforts (optional). The study is based on the logic model that this professional development will change kindergarten pedagogical practices, which in turn will increase and improve children's opportunities for movement, play and exploration, and lead to positive child developmental effects. Thus, the main aim of the professional development is to provide kindergarten staff the necessary expertise and resources to intervene on the child level. Researchers will not directly take part in the delivery of the intervention on the child level. The intervention at the child level is derived from hypotheses, theory and evidence relating to the beneficial effects of movement, play and exploration on children's physical, socio-emotional, and cognitive development. By developing the move-play-explore nexus, the project is transdisciplinary in trying in overcome boundaries between public health, early years pedagogy and movement sciences. The intervention will be delivered by the kindergarten staff through the use of a wide specter of types of activities and play; from child-initiated and directed free-play at the one end, to guided play, and structured teacher-led activities at the other end.

The study will be conducted from August 2024 to June 2026, for which the intervention is adjusted based on a pilot study conducted 2023-2024. Data collection will be performed at baseline (all outcomes), 7-month follow-up (selected outcomes) and 18-month follow-up (all outcomes). In addition, process evaluation measures will be taken throughout the study. Derived from a conservative sample size calculation using standard formulas, including correction for the cluster RCT design, we aim to recruit a minimum of 50 kindergartens and 500 children to the study. This sample size will allow for uncovering statistical significant standardized effect sizes (Cohen's d) of 0.25-0.40.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a participating kindergarten
* Born in 2020

Exclusion Criteria:

* None

Ages: 4 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Movement competence and creativity | Change to 18 months
  The Test of Movement Competence and Creativity, consists of 3 standardized, multi-item movement challenges children will solve as successful or not. Measured as scores.
Movement competence and creativity | Change to 7 months
  The Test of Movement Competence and Creativity, consists of 3 standardized, multi-item movement challenges children will solve as successful or not. Measured as scores.

SECONDARY OUTCOMES:
Physical activity and sedentary time | Change to 18 months
  7-day monitoring Actigraph GT3X+. Measured in average cpm and min/day in intensity zones.
Physical activity and sedentary time | Change to 7 months
  7-day monitoring Actigraph GT3X+. Measured in average cpm and min/day in intensity zones.
Standing long-jump | Change to 18 months
  PREFIT test battery, measured in meters.
Grip strength | Change to 18 months
  PREFIT test battery, measured in kg.
Supine timed up and go | Change to 18 months
  SUNRISE test battery, measured in seconds.
Body mass | Change to 18 months
  Measured in kg.
Body mass index | Change to 18 months
  Measured i kg/meter2.
Children's social-emotional health | Change to 18 months
  The Strength and Difficulties Questionnaire, staff-report on 25 items. Measured as scores.
Behavioural self-regulation | Change to 18 months
  Head-Toes-Knees-Shoulders task (HTKS). Measured as scores.
Numeracy | Change to 18 months
  Early Years Toolbox Numbers task. Measured as scores.
Vocabulary | Change to 18 months
  Early Years Toolbox Vocabulary task. Measured as scores.
Playfulness, explorative behaviour and wellbeing | Change to 18 months
  The Children's Involvement and Wellbeing in Movement, Play and Exploration Questionnaire, staff-report on 21 items. Measured as scores

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Aadland, PhD, Principal Investigator — Western Norway University of Applied Sciences
Locations (1):
- Western Norway University of Applied Sciences, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Data may be shared on reasonable request

REFERENCES:
- [Derived] Aadland E, Sadownik AR, Rudd J, Tjomsland HE, Okely AD, Eriksen PB, Grindheim M, Joyce T, Tveten K, Varnes TK, Johannessen K, Aadland KN, Odegaard EE. Move-play-explore in early childhood education (MoveEarly) - study protocol of a cluster randomized controlled trial of staff professional development for quality pedagogical practices and holistic child development in Norwegian kindergartens. BMC Public Health. 2025 Dec 10;26(1):546. doi: 10.1186/s12889-025-25831-1. PMID 41372827
- See also: Project web page — https://www.hvl.no/en/research/project/moveearly/